CLINICAL TRIAL: NCT04641715
Title: OAGB-MGB Conversion for Failed Procedure: a Multicenter Italian Study
Brief Title: OAGB-MGB Conversions for Post-operative Complications
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Mario Musella MD, Full Professor, Federico II University
Other Study IDs: MGB Class
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: OAGB-MGB — One Anastomosis Gastric Bypass - Mini Gastric Bypass as both restrictive and malabsorptive bariatric procedure

SUMMARY:
Laparoscopic mini/one anastomosis gastric bypass (MGB/OAGB) is a relatively new bariatric procedure and is gaining ground over the surgical approach for morbid obesity as a safe and effective operation. Revision of MGB/OAGB was never studied before as multicenter data collection: we collected data from 21 italian centers who perform MGB/OAGB to evaluate patients' conditions which determinated the conversion from this procedure to another kind of bariatric technique.

DETAILED DESCRIPTION:
MGB / OAGB has been shown to be an effective and safe bariatric technique. Despite that, the complications of this procedure have already been extensively described in the literature. Our goal is to collect data from 21 Italian centers that practice MGB / OAGB to evaluate the reasons and complications that led surgeons to revise this surgery with a subsequent bariatric procedure. For this reason we have analyzed the data provided by the centers on 8676 patients undergoing MGB / OAGB, focusing attention on phenomena such as GERD, anastomotic stenosis, bleeding and marginal ulcers which are the most frequent causes of re-intervention. We also evaluated the changes in BMI between the primary procedure and the revision procedure to ensure that the bariatric purpose of the surgical program was maintained.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent to OAGB-MGB who needed conversion to other bariatric procedure

Exclusion Criteria:

* Patients underwent to OAGB-MGB who needed conversion to other bariatric procedure in emergency within 48/72 hours after the first surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients elegible for conversion from OAGB-MGB to other bariatric procedures
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
Reasons for Conversion from MGB/OAGB to other bariatric procedures | From 2006 to 2020
  We evaluated the reasons for conversion from MGB/OAGB in terms of late post-operative complications.
Surgical type of conversion from MGB/OAGB | From 2006 to 2020
  We evaluated the type of bariatric revisional procedure performed in each patient underwent to MGB/OAGB

CONTACTS AND LOCATIONS:
Overall Officials: Mario Musella, Full Professor, Principal Investigator — Federico II University
Locations (1):
- Nunzio Velotti, Naples, Italy

IPD SHARING:
Plan to Share IPD: No